CLINICAL TRIAL: NCT00802269
Title: Pain Using Reduced Fluence Parameters in Photocoagulation for Diabetic Retinopathy.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-032
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; Laser photocoagulation; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced Fluence Parameters (Experimental): Eyes receiving retinal photocoagulation with reduced fluence parameters (time 20-50 msec, power 400-700 mW)
  Interventions: Procedure: Retinal laser photocoagulation
- Traditional parameters (Active Comparator): Eyes receiving retinal photocoagulation with traditional parameters (time 100-200 msec, power 200-400 mW)
  Interventions: Procedure: Retinal laser photocoagulation

INTERVENTIONS:
Procedure: Retinal laser photocoagulation — Retinal laser photocoagulation using a 532 nm laser
  Other Names: Alcon Eyelite 532 (doubled frequency Nd:Yag)

SUMMARY:
The used of reduced fluence parameters for panretinal photocoagulation decreases pain as perceived by the patient, compared to traditional parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older, that signed informed consent
* Proliferative diabetic retinopathy with indication for panretinal photocoagulation

Exclusion Criteria:

* Previous retinal photocoagulation
* Previous ocular surgical procedures
* Ocular media opacities
* History of trigeminal neuralgia
* Chronic ocular pain
* Depression under conductual or medical treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pain (NRS-11 scale) | Immediately post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Alvarez-Verduzco, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico